CLINICAL TRIAL: NCT06941571
Title: Effect of Solutions Used in Burn Wound Irrigation on Healing, Pain, Fear and Anxiety: Randomized Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nurdan AKCAY DİDİSEN (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor-Investigator, Nurdan AKCAY DİDİSEN, Assoc. Prof., Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20.07.2023/1117; 42497 (Other Grant/Funding Number: Health Institutes of Türkiye)
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Burn; Burn Wound; Healing; Pain; Anxiety; Fear
MeSH Terms: conditions — Burns; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Before data collection, the materials required for the intervention will first be provided. A preliminary application phase will be carried out with six more children. After the use of the data collection tools after the preliminary application, a pre-test measurement will be made for the intervention groups, photographs will be taken and a wound swab sample will be taken. After this shooting, the burn wound will be irrigated and the wound will be covered with a hydrophilic dressing. Three days after the intervention, the children will be called for dressing again. The burn wound will be photographed again and a wound swab sample will be taken. Irrigation will be applied again. With this monitoring, the children will be monitored for 12 days with regular appointments, four times. In the final phase, the burn areas whose photographs were taken will be sent to specialists and they will be asked to make burn area evaluations using the Bates-Jansen wound assessment form.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Burn intervention will be performed by the burn clinic nurse. In this project, the participants who will receive burn dressing, the project manager, project researchers and the statistician who will evaluate the study results will remain blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): In this group, burn wounds will be washed with irrigation solution in accordance with the clinical care protocol (%0.09 NaCl).
- Active Comparator 1 (Active Comparator): In this group, burn wounds will be washed with hypochlorous acid irrigation solution.
  Interventions: Other: Irrigation Solution
- Active Comparator 2 (Active Comparator): In this group, burn wounds will be washed with chlorhexidine gluconate irrigation solution.
  Interventions: Other: Irrigation Solution

INTERVENTIONS:
Other: Irrigation Solution — In this group, the effects of washing burn wounds with different irrigation solutions will be investigated.
  Arms: Active Comparator 1; Active Comparator 2

SUMMARY:
Burn, skin and/or subcutaneous tissues; It is an acute injury that causes traumatic lesions by exposure to thermal, chemical, mechanical or electrical agents. Among all traumatic injuries, burns are the most common type of injury and affect the entire body system. The World Health Organization reports that approximately 180,00 deaths per year are due to burns, making it the fifth most common type of childhood injury. It is also stated that 80% of burned children have hot water burns. Treatment is in two ways: surgical and non-surgical. The type of burn, its size, depth and the individual characteristics of the child affect the type of treatment.

Non-surgical treatment is always the first choice in burn treatment. The primary method of this method is burn dressings. Before dressing, the burn surface must be cleaned/irrigated with an appropriate antiseptic solution to remove metabolic wastes and tissue exudate. The aim here is to prepare a suitable environment for the burn wound to heal and to accelerate the healing process. In the literature, it is recommended to use various antiseptic solutions such as 0.9% NaCl, 0.5% chlorhexidine and hypochlorous acid for irrigation of burn wounds. Applying these solutions involves physical contact with the wound, and this contact may cause pain in the child. Additionally, the temperature and pH of the solution may cause discomfort. The pain that occurs during the irrigation process can further intensify anxiety and fear. However, it is not known which burn solutions used cause more pain, anxiety and fear. In this project, the effects of irrigation solutions used in the care of pediatric burn wounds on pain, fear, anxiety, infection development and healing will be examined. Child patients aged 5-10 years old with limb burns who present with hot water burns and do not have an indication for hospitalization will be included in the project. Children coming to burn dressing will be divided into three groups by simple randomization method. The burn wound of children in the first group will be irrigated with 0.09% NaCl, the children in the second group will be irrigated with 0.5% chlorhexidine, and the burn wound of children in the third group will be irrigated with hypochlorous acid solution. During irrigation of the burn wound, the child's anxiety, fear and pain status will be evaluated. At the same time, the effectiveness of the irrigation solutions used on the development of infection on the wound and its effectiveness on healing will be examined. For this reason, the burn wound will be monitored every three days. For this reason, children will be called to the burn clinic for dressing every three days. Before each dressing, a wound swab sample will be taken to determine the infection status in the burn wound. The Bates-Jensen wound assessment tool will be used to determine the healing status of the burn wound, and this tool will be evaluated by the burn nurse and two pediatric surgeons. In total, children will be monitored for 12 days. At the end of the project, the effect of the solutions used in burn irrigation on infection and healing will be determined. At the same time, the effects of the solutions on anxiety, fear and pain in children will be evaluated. It is thought that the data obtained as a result of the project will contribute to the development of a burn wound care protocol.

DETAILED DESCRIPTION:
Irrigation, debridement and cleaning constitute the basis of standard burn care in wound cleaning. Debridement and wound irrigation/cleaning are critical for the removal of debris and the reduction or elimination of biofilms (Wilkins and Unverdorben, 2013). In an in vitro study on the effectiveness of wound irrigation/cleaning solutions, the importance of measuring protein concentrations on the wound for the effectiveness of solution cleaning is emphasized (Klasinc et al., 2018). It was determined that HOCl solution used in infected wound care irrigation was effective in reducing the number of bacteria in the wound, wound pain, odor, discharge and wound healing (Ragab and Kamal, 2017). In another study on the effect of HOCl solutions, significant reductions in treatment costs were determined due to its contribution to the prevention of biofilm and the acceleration of tissue healing in the wound (Bongiovanni et al., 2016). In another study conducted on patients using 0.9% normal saline and 10% povidone-iodine for irrigation during the wound healing process, it was determined that 5% infection developed after 0.9% normal saline irrigation and 12% infection developed after 10% povidone-iodine irrigation (Kurnia, Widiasih, Rahayu, 2022). In a randomized controlled trial investigating the effectiveness of debridement and wound cleaning with 2% hydrogen peroxide in graft harvesting in chronically colonized burn wounds, grafting was performed after washing the right extremity with 2% hydrogen peroxide gauze for five minutes and normal saline irrigation, and debridement and skin grafting were applied with the conventional method in left extremity wounds. It was found that hydrogen peroxide application was safe and significantly increased the average graft harvesting success rate in chronically colonized wounds (Mohammadi et al., 2013). In another study on the effectiveness of chlorhexidine gluconate in burn wound irrigation/cleaning, it was determined that chlorhexidine was effective against multidrug-resistant organisms (Miller-Willis, Thomas, Joe, 2020). In the project, a culture sample will be taken before irrigation of the burn wound to determine the status of bacterial invasion on the wound. Thus, the effectiveness of the solutions used against bacterial organisms will be determined. At the same time, the healing status of the burn wound will be determined in terms of size, depth, edges, tunneling, type and amount of necrotic tissue, type and amount of exudate, color of the skin around the wound, peripheral tissue edema and edema, granulation tissue and epithelialization with the Bates-Jensen wound assessment tool, which will be evaluated by a burn nurse and two pediatric surgeons who are actively working in the field. In childhood burns, pain, medical procedures, and long-term treatment protocols after the injury process also cause a series of psychological and physical reactions in children. Therefore, burns are one of the most traumatic injuries a child can experience (Wickens et al., 2023). Therefore, acute pain, anxiety, and fear management must be provided during dressing changes in children and must be controlled with a child-centered approach. In another study conducted on the relationship between pre-procedure anxiety and procedure-related pain during outpatient pediatric burn care, more than half of the patients were found to have mild anxiety and approximately 5% of the patients had severe anxiety. The study also reported that younger children (6-8 years old) had higher anxiety scores than older children (15-17 years old). It was also found that anxiety before dressing changes in outpatient pediatric burn patients was significantly associated with self-reported general moderate-severe pain (Vest et al., 2023; Zhang et al., 2020). In another study investigating the effect of desktop virtual reality on pain and anxiety during burn wound cleaning/debridement in infants and young children, it was found that six-year-old children experienced severe pain during 10 minutes of burn wound cleaning (Alrimy et al., 2023). Although pharmacological and non-pharmacological treatments have developed in the burn care approach today, the management of acute pain, anxiety and fear in children is among the situations encountered during care protocols. When this situation is not evaluated with an appropriate approach with symptom controls, it can cause long-term negative effects on children. In particular, in the literature, anxiety-fear and anxiety are considered as two important factors causing procedural pain due to dressing changes. In addition, it has been emphasized that negative pain experiences during procedural interventions can have lifelong effects on children. Therefore, in the pediatric approach, it is an important issue not only to treat the child's pain, but also to treat acute pain and anxiety due to debridement and dressing changes. In outpatient settings, non-pharmacological distraction and comfort methods such as benzodiazepines, ketamine, oral opioids and topical lidocaine are frequently used (Hansen et al., 2019). In a study conducted to examine the wound care practices of nurses working in a university hospital, it was determined that 45.1% of the nurses applied analgesics if requested by the doctor, and 29.7% did not routinely apply analgesics before dressing during dressing application (Rızalar et al., 2019). Solutions used in burn wound irrigation in children may cause pain due to physical pain and sensitivity; the temperature and pH level of the solution may also cause discomfort. Psychological effects are also important; children may often experience fear and anxiety in the hospital environment and during medical interventions. Therefore, health professionals should be careful to closely monitor, observe and record the characteristics of the wound, and pay attention not only to the wound but also to the changing facial expressions during dressing in order to consider the patient as a whole. In conclusion, there are several gaps in current burn wound irrigation treatment. The inconsistency of methods and solutions used in different clinics and countries leads to differences in treatment outcomes. Problems such as the lack of a clear consensus in the selection of antiseptics and cleansers, effective management of pain and anxiety in children, inadequacy of current methods in infection control and side effects of solutions are prominent. In addition, accessibility and cost issues of treatment materials in low- and middle-income countries, lack of knowledge of health professionals and lack of standardized protocols also negatively affect the quality of treatment. More research, standardization, education and accessibility of resources are important to eliminate these gaps.

ELIGIBILITY:
Inclusion Criteria: The child must be between the ages of 5-10, be followed up in the burn clinic of the pediatric surgery service, be conscious, alert, and open to communication, be a child with 10% or 2nd degree superficial and deep burns who are being followed up as an outpatient, have burns on the arms, legs, and torso, have hot water (boiling water, etc.) burns, and the parent and child must agree to participate in the study.

Exclusion Criteria: The child must be younger than 5 years old or older than 10 years old, have a general condition disorder due to burns, have a change in consciousness, have genital area and facial burns, have a 10% or more second and third degree burn, have a burn that is an indication for hospitalization, the parent uses topical agents for burn healing at home, and the parent and child do not accept to participate in the study.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker Facial Expression Rating Scale Score | 4 months
  The effects of different irrigation solutions on pain will be measured.
Child Fear Scale Score | 4 months
  The effects of different irrigation solutions on fear will be measured..
Child State Anxiety Scale Score | 4 months
  The effects of different irrigation solutions on anxiety will be measured..

IPD SHARING:
Plan to Share IPD: No